CLINICAL TRIAL: NCT07018544
Title: A Multicentre, Prospective, Single-arm, Non-interventional Regulatory Post-marketing Surveillance (rPMS) Study to Investigate the Safety and Effectiveness of Wegovy® (Semaglutide) in Patients With Obesity and Patients With Overweight in Routine Clinical Practice in Korea.
Status: Enrolling by invitation | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9536-7543; U1111-1281-9419 (Other: WHO)
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Obesity and Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — semaglutide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Semaglutide: Participants will be treated with commercially available semaglutide according to the approved label and to real-world clinical practice at the discretion of the treating physician. The decision to treat participants with semaglutide has been made by the treating physician independently from the decision to include the participants in this study.
  Interventions: Other: semaglutide

INTERVENTIONS:
Other: semaglutide — Participants will be treated with commercially available semaglutide according to routine clinical practice at the discretion of the treating physician.
  Other Names: Wegovy

SUMMARY:
This study is conducted to investigate the safety and effectiveness of semaglutide in participants with obesity and overweight in routine clinical practice. Participants will get semaglutide as prescribed by a doctor. This study will last for about 4 years and participants will participate in the study for approximately 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
2. The decision to initiate treatment with commercially available semaglutide has been made by the participants and the treating physician before and independently from the decision to include the participant in this study.
3. Male or female adults, age above or equal to 19 years who is scheduled to start treatment with semaglutide based on the clinical judgment of their treating physician as specified in the Korean-prescribing Information (approved label in Korea) at the time of signing informed consent.

Exclusion Criteria:

1. Participants who are or have previously been on semaglutide therapy before enrollment.
2. Known or suspected hypersensitivity to the active substance or any of the excipients of semaglutide.
3. Previous participation in this study. Participation is defined as having given informed consent in this study.
4. Female participant who is pregnant, breast-feeding, or intends to become pregnant and is of childbearing potential not using adequate contraceptive methods (adequate contraceptive measures as required by local regulation or practice).
5. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will be treated with commercially available semaglutide according to the approved label and to real-world clinical practice at the discretion of the treating physician. The decision to treat participants with semaglutide has been made by the treating physician independently from the decision to include the participants in this study.
Sampling Method: Non-Probability Sample
Enrollment: 840 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Number (incidence) of AEs | From Visit 1 (baseline, 0 week) to Visit 4 (22 weeks < ~ ≤ 30 weeks)
  Count of events

SECONDARY OUTCOMES:
Number (incidence) of ADRs | From Visit 1 (baseline, 0 week) to Visit 4 (22 weeks < ~ ≤ 30 weeks)
  Count of events
Number (incidence) of SAEs | From Visit 1 (baseline, 0 week) to Visit 4 (22 weeks < ~ ≤ 30 weeks)
  Count of events
Number (incidence) of SADRs | From Visit 1 (baseline, 0 week) to Visit 4 (22 weeks < ~ ≤ 30 weeks)
  Count of events
Number (incidence) of unexpected AEs | From Visit 1 (baseline, 0 week) to Visit 4 (22 weeks < ~ ≤ 30 weeks)
  Count of events
Number (incidence) of unexpected ADRs | From Visit 1 (baseline, 0 week) to Visit 4 (22 weeks < ~ ≤ 30 weeks)
  Count of events
Number (incidence) of unexpected SAEs | From Visit 1 (baseline, 0 week) to Visit 4 (22 weeks < ~ ≤ 30 weeks)
  Count of events
Number (incidence) of unexpected SADRs | From Visit 1 (baseline, 0 week) to Visit 4 (22 weeks < ~ ≤ 30 weeks)
  Count of events
Total dose of semaglutide | From Visit 1 (baseline, 0 week) to Visit 4 (22 weeks < ~ ≤ 30 weeks)
  Milligram/milliliter (mg/mL)
Body weight loss | From Visit 1 (baseline, 0 week) to Visit 4 (22 weeks < ~ ≤ 30 weeks)
  Percent (%)
Body weight loss | From Visit 1 (baseline, 0 week) to Visit 4 (22 weeks < ~ ≤ 30 weeks)
  Kilogram (kg)
The proportion of participants losing greater than or equal to 5% body weight | From Visit 1 (baseline, 0 week) to Visit 4 (22 weeks < ~ ≤ 30 weeks)
  Percent (%)
The proportion of participants losing greater than or equal to 10% body weight | From Visit 1 (baseline, 0 week) to Visit 4 (22 weeks < ~ ≤ 30 weeks)
  Percent (%)
The proportion of participants losing greater than or equal to 15% body weight | From Visit 1 (baseline, 0 week) to Visit 4 (22 weeks < ~ ≤ 30 weeks)
  Percent (%)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (8):
- South Korea (8):
  - MyongJi Hospital, Goyang-si, Gyeonggi-do
  - Kosin University Gospel Hospital, Busan
  - Yonsei Hanaro Clinic, Chungcheongnam-do
  - Daejeon Endo Internal Medicine Clinic, Daejeon
  - Ajou University Hospital, Gyeonggi-do
  - Samsung Medical Center, Seoul
  - Hplus Yangji Hospital, Seoul
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com